CLINICAL TRIAL: NCT03155529
Title: Three-dimensional Study on the Structural Destruction of Pelvic Organs and Pelvic Floor After Radical Hysterectomy in Cervical Cancer
Brief Title: Three-dimensional Study on the Structural Destruction of Pelvic Anatomy in Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Sponsor
Other Study IDs: NFEC2013032-0
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2016-09

CONDITIONS: Cervical Cancer; Postoperative Pelvic Floor Dysfunction
Keywords: cervical cancer; radical hysterectomy; Postoperative pelvic floor dysfunction; the injure of pelvic floor; Three-dimensional reconstruction; structural destruction of pelvic organs; structural destruction of pelvoic floor
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- radical hysterectomy group: Using dynamic MRI and 3D reconstruction to assess the effect of RH on pelvic floor muscles and pelvic organs (location and mobility of bladder neck and urethral).
  Inclusion Criteria： ①Patients diagnosed as FIGO stage IA2、IB1、IIA1 cervical cancer ; ②Patients diagnosed as FIGO stage IB2、IIA2 cervical cancer, eligible for RH after neoadjuvant chemotherapy; ③Patients diagnosed as FIGO stage IIA endometrial carcinoma; ④Patients didn't have pelvic organ prolapse and urinary incontinence; ⑤Ability to hold Valsalva for dynamic MRI; ⑥Patients aged 20-70 years; ⑦Patients undergone RH surgery; ⑧Informed consent was signed.
  Exclusion Criteria：
  ①With MRI or urodynamic examination contraindication; ②Previously undergone POP or SUI surgery; ③BMI>30 ④With serious postoperative complications.
  Interventions: Procedure: radical hysterectomy

INTERVENTIONS:
Procedure: radical hysterectomy — A standard radical hysterectomy with lymphadenectomy was performed. Static and dynamic MRI were performed. A suggested urodynamic examination was done according to the ICS. A 3D reconstruction technique was used to construct the 3D model of the pelvis, pelvic floor muscle, pelvic organ such as bladder and urethral.

SUMMARY:
Cervical cancer is one of the most prevalent malignancies in female .To the younger patients, radical hysterectomy which is a standard operation during the earlier and middle therapy stage as well as more effective technique like radiotherapy and chemotherapy give them a longer life expectancy. However, the operation destroys patients' normal pelvic anatomy, nutrient supplements and internal secretion so that postoperative pelvic floor functional dysfunction has a destructive effect for their life. There are tremendous studies on clinical symptoms while few on anatomical changes and the relationship between pelvic floor symptoms and the dysfunction. Two-dimensional Magnetic Resonance Imaging(MRI), transperineal ultrasonography， Urodynamic examination and anorectal manometry are frequently used in the fine-structure varies and pelvic floor function. Now three-dimensional MRI has more advantages in fine change of Pelvic anatomical and space position，as well as clearly showing the relationships between the change and space with the pelvic floor function. Based on an eight-year-study on three-dimensional MRI, we can analyze the postoperational anatomical changes and the relationship between the changes and the dysfunction by combined anatomic parameters which are measured on static-dynamic three- dimensional model with clinical symptoms, transperineal ultrasonography,urodynamic examination and anorectal manometry. We expect our study could provide scientific basis for on protective and repaired measures of pelvic floor.

ELIGIBILITY:
Inclusion Criteria： ①Patients diagnosed as FIGO stage IA2、IB1、IIA1 cervical cancer ; ②Patients diagnosed as FIGO stage IB2、IIA2 cervical cancer, eligible for RH after neoadjuvant chemotherapy; ③Patients diagnosed as FIGO stage IIA endometrial carcinoma; ④Patients didn't have pelvic organ prolapse and urinary incontinence; ⑤Ability to hold Valsalva for dynamic MRI; ⑥Patients aged 20-70 years; ⑦Patients undergone RH surgery; ⑧Informed consent was signed.

Exclusion Criteria：

①With MRI or urodynamic examination contraindication; ②Previously undergone POP or SUI surgery; ③BMI>30 With serious postoperative complications.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a study comparing 70 cases (cervical cancer patients before RH surgery) to 70 controls (Same group cervical cancer patients before RH surgery) exams.All recruits will undergo the MRI evaluation,transperineal ultrasonography, urodynamic examination and anorectal manometryand the basic information of them will be recorded.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
levator ani muscle space coordinates. | september 3,2017 to september 1,2019

SECONDARY OUTCOMES:
Bladder，uterus and rectum space coordinates. | september 3,2017 to september 1,2019

OTHER OUTCOMES:
bladder neck, internal cervix, external cervix, anorectal junction's distance from the PCL line | september 3,2017 to september 1,2019
levator hiatus width and length, Levator symphasis gap leftside and rightside,levator plate angle. | september 3,2017 to september 1,2019
Urethral rotation Angle,posterior vesicourethral angle. | september 3,2017 to september 1,2019

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No